CLINICAL TRIAL: NCT04719078
Title: Prospective Assessment of MRI for Morphological and Functional Imaging in the Thorax.
Brief Title: Thorax MRI for Evaluation of Lung Morphology, Ventilation and Perfusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MR 02
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Lung Diseases; Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases; Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: Prospective, single-centre, non-randomised, non-blinded trial with MR-Imaging of patients. All of the patients undergo MR-Imaging as well as the two standard diagnostic procedures: CT and lung function tests.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Other): There are no study arms. All patients obtain all imaging modalities.
  Interventions: Diagnostic Test: MRI of the chest

INTERVENTIONS:
Diagnostic Test: MRI of the chest — The study participants will obtain a MRI of the thorax with one of the institutions MR machines (Philips Achieva 1.5T, GE Discovery 3T, MRI Siemens Skyra 3T, and GE SIGNA Artist 1.5T). The study participant will be asked to lie in the MR scanner for about 30 minutes while the images will be acquired. The image acquisition with the above-mentioned MR machines is authorised in Switzerland and the application is done according to the product information.

SUMMARY:
In spite of the considerable technical difficulties, several publications confirm the potential that T1-maps and MRI to characterize pathological changes in lung tissue. However, existing literature still cannot provide a final evaluation of the presented methods. Study participants won't have any disadvantage in participating the study since all of them undergo next to the MRI-Scan also the two standard methods: CT and lung function test.

In this study the value of chest MR compared to CT and LFT in the evaluation of morphological lung changes and their correlation to lung ventilation and perfusion will be evaluated.

DETAILED DESCRIPTION:
Patients with interstitial lung disease require an adequate tool for diagnosis and monitoring. Traditionally, the diagnostics are done by CT and lung-function tests. Follow-up of these patients include regular CT-Imaging and LFT to monitor disease progress to visualize possible complications early. Every examination exposes the patient to ionizing radiation, and LFTs alone are not sensitive enough to visualize local changes. Therefore, it is desirable to switch from these two diagnostic tools to a less harm-full and a more sensitive one: MR-Imaging. MR-Imaging allows for a non-invasive and more sensitive illustration of lung morphology as well as local ventilation and perfusion for early detection of lung function alterations without the exposure of the patient to ionizing radiation.

1. Ojective To demonstrate the value of MR-Imaging as a valuable, radiation-free method to visualize lung morphology and pathologic lung changes in patients with interstitial lung diseases quantitatively and qualitatively. A positive result would allow using MR as an additive or alternative method in the assessment of parenchymal lung changes to detect early parenchymal changes as well as to monitor the course of disease, especially for medical treatment.
2. Objective Quantitative and qualitative validation of MR-Imaging in the assessment of local lung ventilation and perfusion compared to lung function tests.

Prospective, single-centre, non-randomised, non-blinded trial with MR-Imaging of patients. All of the patients undergo MR-Imaging as well as the two standard diagnostic procedures: CT and lung function tests.

Inclusion criteria: patients with interstitial lung disease scheduled for CT and LFT, written consent, ≥ 18 years.

Exclusion criteria: claustrophobia and impossibility to lie in the MR for more than 30 minutes, pregnancy, and the generally valid contraindications for MRI.

The study participants will obtain a MRI of the thorax with one of the institutions MR machines (Philips Achieva 1.5T, GE Discovery 3T, MRI Siemens Skyra 3T, and GE SIGNA Artist 1.5T). The study participant will be asked to lie in the MR scanner for about 30 minutes while the images will be acquired. The image acquisition with the above-mentioned MR machines is authorised in Switzerland and the application is done according to the product information.

ELIGIBILITY:
Inclusion Criteria:

* patients with interstitial lung disease scheduled for CT and LFT
* written consent
* ≥ 18 years.

Exclusion Criteria:

* claustrophobia
* impossibility to lie in the MR for more than 30 minutes
* pregnancy
* generally valid contraindications for MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Lung Morphology | 2 years
  Value of static MR-images compared to CT.

SECONDARY OUTCOMES:
Lung function | 2 years
  Correlation of functional MR with lung function ventilation/perfusion compared to CT.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich - Diagnostic Radiology, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No